CLINICAL TRIAL: NCT06342791
Title: Effect of Laser Acupuncture on Menstrual Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Ali Galal El Sayed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 004349
Record Dates: First submitted 2024-02-14; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Laser Acupuncture; Low Back Pain; Menstruation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: two groups
Who Masked: Participant
Masking Description: laser acupuncture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (study group) (Experimental): received Laser on acupuncture point BL23, BL26, BL40, SP6
  Interventions: Device: laser acupuncture
- Group B (Control group) (Placebo Comparator): received sham laser acupuncture on BL23, BL26, BL40, SP6 but the laser was not turned on
  Interventions: Device: laser acupuncture

INTERVENTIONS:
Device: laser acupuncture — laser use to stimulate acupuncture points

SUMMARY:
effect of laser acupuncture on menstrual back pain

DETAILED DESCRIPTION:
The aim of this study is to determine the effect of laser acupuncture on the points BL23, BL26, BL40 and SP6 in relieving menstrual back pain.

ELIGIBILITY:
Inclusion Criteria:

* All females will have low back pain during menstruation
* Age of the patients will range from 20-30 years.
* Their BMI will be range from 20-30 kg/ m 2

Exclusion Criteria:

* - Psychiatric disorders
* Pelvic floor dysfunction
* Lumber disc prolapse or any Previous surgery on spine.
* Tumor in lumbar spine

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — - Female who suffers from low back pain during menstruation.
Enrollment: 32 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-05-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
back Pain intensity during menstruation | before 3 month from begining of treatment
  It will be assess by Visual analogue scale(VAS). VAS used to indicate the level of pain intensity from 1 to 10, before starting treatment (first record) then after treatment (as second record). A visual analogue scale's (VAS) baseline typically falls at one end of the scale and is frequently denoted by the numbers "no pain" or "0," which indicate for the absence of the sensation being assessed. The other end of the line indicates "worst pain imaginable" or a high numerical value, such as 10
pain threshold | Before 3 month from begining of the treatment
  Using algometer to measure pain threshold. Before beginning the measurement, a pressure algometer's baseline is usually set at zero pressure. This means that the initial pressure applied by the algometer is zero, and then the pressure is gradually increased until the individual being tested starts to feel pain or discomfort. This baseline helps to establish a reference point for measuring pain thresholds or sensitivity to pressure
Ability to perform daily activities | Before 3 month from begining of the treatment
  Ability to perform daily activities will be assess by using Instrumental activities of daily living (IADL).This scale has been designed to give information about how back pain has affected the ability to manage everyday life. IADLs are scored based on what an individual can do rather than what she is doing. Ask patient to answer every section and mark in each section only the one box which most closely describes the condition at this time. There are 22 questions and rate them on the scale at right. The higher scores mean a better.

SECONDARY OUTCOMES:
back Pain intensity during menstruation | 3 month after treatment
  It will be assess by Visual analogue scale(VAS). VAS used to indicate the level of pain intensity from 1 to 10, before starting treatment (first record) then after treatment (as second record). A visual analogue scale's (VAS) baseline typically falls at one end of the scale and is frequently denoted by the numbers "no pain" or "0," which indicate for the absence of the sensation being assessed. The other end of the line indicates "worst pain imaginable" or a high numerical value, such as 10
pain threshold | 3 month after treatment
  Using algometer to measure pain threshold. Before beginning the measurement, a pressure algometer's baseline is usually set at zero pressure. This means that the initial pressure applied by the algometer is zero, and then the pressure is gradually increased until the individual being tested starts to feel pain or discomfort. This baseline helps to establish a reference point for measuring pain thresholds or sensitivity to pressure
Ability to perform daily activities | 3 month after treatment
  Ability to perform daily activities will be assess by using Instrumental activities of daily living (IADL).This scale has been designed to give information about how back pain has affected the ability to manage everyday life. IADLs are scored based on what an individual can do rather than what she is doing. Ask patient to answer every section and mark in each section only the one box which most closely describes the condition at this time. There are 22 questions and rate them on the scale at right. The higher scores mean a better.

CONTACTS AND LOCATIONS:
Overall Officials: Cairo University, Principal Investigator — Faculty of physical therapy cairo universty
Locations (1):
- Faculty of physical therapy cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and informed consent form
Supporting Information: Study Protocol, ICF
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research. and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).